CLINICAL TRIAL: NCT05891873
Title: Delirium in the (Neuro)Intensive/Critical Care in the Adult and Paediatric Czech Populations
Status: Recruiting | Type: Observational
Sponsor: Masaryk University (Other)
Collaborators: Brno University Hospital (Other); University Hospital, Motol (Other)
Responsible Party: Sponsor
Other Study IDs: DELUSION-DEEP-CZ
Record Dates: First submitted 2023-05-17; First posted 2023-06-07 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Delirium
Keywords: delirium; delirium screening; ICU delirium
MeSH Terms: conditions — Delirium | interventions — Electroencephalography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Neurointensive/neurocritical group (N-ICU)
  Interventions: Diagnostic Test: CAM-ICU; Diagnostic Test: ICDSC; Diagnostic Test: 4AT; Diagnostic Test: MASTcz (The Mississippi Aphasia Screening Test); Diagnostic Test: EEG
- Paediatric intensive/critical group (P-ICU)
  Interventions: Diagnostic Test: p(s)CAM-ICU; Diagnostic Test: CAPD; Diagnostic Test: EEG

INTERVENTIONS:
Diagnostic Test: CAM-ICU — Patients who meet the inclusion criteria will be screened daily for delirium using the screening test mentioned above.
  Groups: Neurointensive/neurocritical group (N-ICU)
Diagnostic Test: ICDSC — Patients who meet the inclusion criteria will be screened daily for delirium using the screening test mentioned above.
  Groups: Neurointensive/neurocritical group (N-ICU)
Diagnostic Test: 4AT — Patients who meet the inclusion criteria will be screened daily for delirium using the screening test mentioned above.
  Groups: Neurointensive/neurocritical group (N-ICU)
Diagnostic Test: p(s)CAM-ICU — Patients who meet the inclusion criteria will be screened daily for delirium using the screening test mentioned above.
  Groups: Paediatric intensive/critical group (P-ICU)
Diagnostic Test: CAPD — Patients who meet the inclusion criteria will be screened daily for delirium using the screening test mentioned above.
  Groups: Paediatric intensive/critical group (P-ICU)
Diagnostic Test: MASTcz (The Mississippi Aphasia Screening Test) — People with aphasia will be examined by a skilled speech therapist.
  Groups: Neurointensive/neurocritical group (N-ICU)
Diagnostic Test: EEG — Patients with positive delirium will undergo EEG examination. 10-min native EEG.

SUMMARY:
Intensive and critical care in the intensive care unit (ICU) is often associated with ICU delirium and post-ICU dementia, regardless of the nature of the primary disease or insult. Optimal practical management of ICU delirium including its screening, prevention, and treatment, is an integral part of the current recommendations for optimal ICU care, but there are large gaps in the knowledge about the optimal and most effective prevention and treatment of this complication. Information on the actual implementation of these recommendations in the Czech Republic is lacking. The diagnosis of delirium is particularly challenging in neurointensive care patients (due to overlap with symptoms of primary brain lesions) and in a paediatric population. A complementary multicentre observational 4-year follow-up study, performed in an adult neurointensive/critical care stroke cohort and in a paediatric intensive/critical care cohort in centres following currently recommended preventive measures (Delusion-deep-cz) will investigate the incidence of ICU delirium and post-ICU dementia and their modifiable and non-modifiable predisposing and precipitating risk factors. Objectives are to determine the optimal methods for diagnostic screening of these complications and for the differential diagnosis of conditions mimicking delirium (non-convulsive epileptic state) or symptoms hindering its diagnosis (aphasia), and to study the association between sleep disturbances and ICU delirium to verify the role of sleep in the pathophysiology of delirium.

DETAILED DESCRIPTION:
Design

• Multicentre observational follow-up cohort study with 2 different cohorts and a minimum follow-up period of 6 months.

Recruitment (groups)

1. Neurointensive/neurocritical group (N-ICU): patients with acute ischaemic or haemorrhagic stroke admitted to the Stroke Unit or ICU of the Department of Neurology, University Hospital Brno (NK-UHB).
2. Paediatric intensive/critical group (P-ICU): children aged 6-18 years, admitted to the Paediatric ICU - Department of Paediatric Anaesthesiology and Intensive Care (KDAR-UHB) with a stay of at least 24 hours (including postoperative care).

General working hypotheses

* Current recommendations for the practical management (PADIS) and prevention of delirium lead to a decrease in the incidence of ICU-delirium and post-ICU dementia and may also change the spectrum of significant risk factors.
* In the Czech Republic, both general knowledge and practical implementation of these recommendations may be low.
* Currently recommended screening instruments for ICU-delirium are valid and reliable in both adult and paediatric cohorts of (neuro)intensive/critical patients and can replace the expert assessment using DSM-IV or V criteria (The Diagnostic and Statistical Manual of Mental Illnesses).
* Non-convulsive status epilepticus (NCSE) may mimic ICU-delirium and a routine EEG exam in patients meeting the criteria for ICU delirium may be helpful.
* Aphasia may complicate the diagnosis of delirium and may prevent the use of the current screening tools for delirium in neurointensive care patients.
* Sleep disturbances in ICU patients are often associated with the development of ICU delirium and evaluating the time course of these conditions may reveal their possible causal relationship.

Outcomes Primary outcomes

* Development of ICU delirium Secondary outcomes
* Length of stay in ICU
* Case-fatality risk
* Post-ICU dementia (BDS, Blessed dementia scale)
* Degree of functional dependency (Barthel index)

Objectives

* To review the incidence and significant modifiable and non-modifiable predisposing and precipitating risk factors for ICU delirium and post-ICU dementia in general and neuro-intensive/critical care in adult and paediatric populations treated in health care facilities according to current recommendations for prevention of these complications (ABCDEF bundle).
* To verify optimal methods for diagnostic screening of ICU delirium: CAM-ICU (The confusion assessment method for the ICU), 4AT (Rapid clinical test for delirium detection - 4AT) and ICDSC (Intensive care delirium screening checklist) in adult populations and pCAM-ICU (paediatric confusion assessment method for the ICU), psCAM-ICU (pre-school confusion assessment method for the ICU) and CAPD (Cornell Assessment of Pediatric Delirium) in paediatric populations to screen for delirium.
* To verify optimal methods for the differential diagnosis of conditions that mimic or complicate the diagnosis of ICU delirium: NCSE, aphasia,
* To investigate associations between sleep disturbances and ICU-delirium to confirm their role in the pathophysiology of delirium.

ELIGIBILITY:
Inclusion Criteria:

* Neurointensive/neurocritical group (N-ICU): patients with acute ischaemic or haemorrhagic stroke admitted to the Stroke Unit or ICU of the Department of Neurology, University Hospital Brno (NK-UHB).
* Paediatric intensive/critical group (P-ICU): children aged 6-18 years, admitted to the Paediatric ICU - Department of Paediatric Anaesthesiology and Intensive Care (KDAR-UHB) with a stay of at least 24 hours (including postoperative care).

Exclusion Criteria:

* (N-ICU) severe trauma with short life expectancy (days)
* duration of the ICU stay shorter than 24 hours

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Neurointensive/neurocritical group (N-ICU): patients with acute ischaemic or haemorrhagic stroke admitted to the Stroke Unit or ICU of the Department of Neurology, University Hospital Brno (NK-UHB).
  Paediatric intensive/critical group (P-ICU): children aged 6-18 years, admitted to the Paediatric ICU - Department of Paediatric Anaesthesiology and Intensive Care (KDAR-UHB) with a stay of at least 24 hours (including postoperative care).
Sampling Method: Non-Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2023-09-07 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants who develop ICU delirium | up to 14 days after admission
  assessed by experienced neuro-intensivist

SECONDARY OUTCOMES:
Length of stay in ICU | up to 10 weeks
Mortality | 6 months
Number of participants and severity of post-ICU dementia, cognitive impairment(Blessed dementia scale, BDS) | 6 months
Degree of functional dependency (Barthel index) | up to 10 weeks and after 6 months
  the higher score, the worse result meaning cognitive impairment and non-independence

CONTACTS AND LOCATIONS:
Locations (1):
- Brno University Hospital, Brno, Czechia

IPD SHARING:
Plan to Share IPD: Undecided